CLINICAL TRIAL: NCT04102709
Title: Spire Medical Health Tag Actigraphy and Sleep Validation in Adults
Status: Completed | Type: Observational
Sponsor: Spire, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-05-16
Record Dates: First submitted 2019-07-24; First posted 2019-09-25 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Health Tag — Health Monitoring Device

SUMMARY:
The purpose of this study is to collect data to validate the step- (actigraphy) and sleep-tracking performance of the Medical Health Tag device developed by Spire Health.

DETAILED DESCRIPTION:
The purpose of this study is to collect data to validate the step- (actigraphy) and sleep-tracking performance of the Medical Health Tag device developed by Spire Health. The step data will be evaluated in a controlled environment over a range of approximately 1.0-2.5 miles per hour (i.e., slow to moderate walking) via Reference manual counting and pedometer. The sleep data will be evaluated in a natural environment (i.e., the participant's daily life and home) over one afternoon and night with Reference sleep/wake data.

ELIGIBILITY:
Inclusion Criteria:

Subject must have the ability to understand and provide written informed consent Subject is over 18 years of age Subject must be willing and able to comply with study procedures and duration Subject is a non-smoker Male or female of any race

Exclusion Criteria:

* Subject is considered as being morbidly obese (defined as BMI >39.5)
* Any medical condition that may prevent successful completion of the tasks in a healthy manner.

  * those requiring a wheelchair or who are housebound (haven't left their home without assistance in the last week)
  * Sleep disorder
  * Gait issue
* Subjects with known respiratory conditions such as severe asthma, flu, bronchitis, or shortness of breath.
* Subjects with self-reported heart or cardiovascular conditions such as congestive heart failure (CHF) or history of stroke or heart attack.
* Any neurological condition such as Parkinson's, Alzheimer's, and Epilepsy
* Subjects experiencing significant sleep impairment or sleep disturbances
* Those with insufficient English language skills to either fully evaluate their understanding of these exclusion criteria during screening or that would otherwise impair their ability to fully participate
* Pregnant at the time of the study
* Unwilling to commit, in writing, to:

  * be on-time for the study
  * be on-time returning the devices the following day
  * avoid alcohol or intoxicants before and during the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subject selection will be a mix of males and females with diverse physiques. Healthy individuals 18 years or older, from the general population will be recruited for participation. The subjects must understand the study and consent to participate by signing the Informed Consent Form. The subjects must be healthy showing no evidence of medical problems as indicated by satisfactorily completing the health assessment form. Eligible subjects need to meet all of the inclusion criteria and none of the exclusion criteria for participation.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2019-09-18 (Actual)

PRIMARY OUTCOMES:
Evaluate the performance of the HT's step algorithm at different walking speeds. | One day
  Accuracy of the Medical Health Tag for the measurement of steps to the Reference
Evaluate the performance of the HT's sleep algorithm accuracy in classifying sleep and wake. | One day
  Accuracy of the HT for the measurement of 60 seconds sleep epochs and total sleep time

CONTACTS AND LOCATIONS:
Overall Officials: Neema Moraveji, Principal Investigator — Chief Scientific Officer
Locations (1):
- Spire, Inc., San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
To be determined.